CLINICAL TRIAL: NCT02455271
Title: Investigation of the Safety and Efficacy of Long Term Administration of Eszopiclone in Insomnia Patients (Study LUN02T)
Brief Title: Investigation of the Safety and Efficacy of Long Term Administration of Eszopiclone in Insomnia Patients
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: LUN02T
Record Dates: First submitted 2015-05-19; First posted 2015-05-27 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2017-01

CONDITIONS: Insomnia
Keywords: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Eszopiclone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with insomnia: Participants with insomnia who will receive eszopiclone per approved label.
  Interventions: Drug: Eszopiclone

INTERVENTIONS:
Drug: Eszopiclone — The usual dosage of eszopiclone is 2 mg per dose for adults and 1 mg per dose for elderly participants, taken orally before bedtime. The dosage may be adjusted according to the participant's symptoms, but a single dose should not exceed 3 mg in adults and 2 mg in elderly participants.
  Other Names: EZOP; Lunesta

SUMMARY:
To investigate the safety and efficacy of administration of eszopiclone for 6 months in insomnia participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have completed LUN01S and need to continue eszopiclone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who have completed Study LUN01S and need to continue eszopiclone
Sampling Method: Non-Probability Sample
Enrollment: 438 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2015-03-30 (Actual); Study Completion 2015-12-22 (Actual)

PRIMARY OUTCOMES:
Assessment of overall improvement | At month 3
  Participants will be interviewed regarding sleep improvement at 3 months after first dose or discontinuation, relative to predose, and select the appropriate answer of: 1. Improved 2. Unchanged 3. Worse 4. Indiscernible
Assessment of overall improvement | At month 6
  Participants will be interviewed regarding sleep improvement at 6 months after first dose or discontinuation, relative to predose, and select the appropriate answer: 1. Improved 2. Unchanged 3. Worse 4. Indiscernible

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Akira Endo, Study Director — Drug Fostering and Evolution Coordination Department, Corporate Medical Affairs Headquarters, Eisai Co., Ltd.
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo

REFERENCES:
- [Result] Japanese Journal of Sleep Medicine 11: 81-94, 2017.